CLINICAL TRIAL: NCT04771338
Title: Examining the Effects of a Job Entry Intervention
Acronym: IMPRESSIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Helen Genova, Associate Director, Center for Autism Research, Kessler Foundation
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R-1078-19
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Autism Spectrum Disorder; Autism; ASD
Keywords: Autism; ASD; Job reentry; Employment intervention; Virtual reality; VR
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Virtual Reality Job Interview Training & character strength training (KF-STRIDE)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Job interview training protocol for 12 sessions
  Interventions: Behavioral: VR-JIT/KF-STRIDE
- Control group (No Intervention): No participation in any intervention protocol

INTERVENTIONS:
Behavioral: VR-JIT/KF-STRIDE — Treatment group will receive 12 sessions of job interview training protocol.
  Other Names: Virtual Interview Training for Transition Age Youth (VIT-TAY); Kessler Foundation STRength IDentification and Expression tool (KF-STRIDE)
  Arms: Treatment group

SUMMARY:
The current study will examine the efficacy of a virtual reality (VR) intervention as well as a newly developed Kessler Foundation STRength IDentification and Expression tool (VR-STRIDE) with adolescents diagnosed with autism spectrum disorder.

DETAILED DESCRIPTION:
The current study will examine the efficacy of a virtual reality (VR) intervention entitled "IMPRoving Expression of Skills and Strengths In Interviewing in a Virtual Environment" (IMPRESSIVE) which targets social competency skills needed for successful job interviewing. Specifically, 2 VR tools are utilized in the IMPRESSIVE intervention. The first tool is VR-Job Interview Training, a VR program which offers the opportunity for repeated practice with a virtual human interviewer. Preliminary evidence suggests that the VRprogram is successful in adults with ASD and schizophrenia in improving interview abilities. However, the efficacy of it has not been evaluated in adolescents with ASD. This represents a significant void in our knowledge, as we do not know whether this program is effective for youth. In addition to VR training, a newly developed tool is included in the currently proposed intervention: the Kessler Foundation STRength IDentification and Expression tool (VR-STRIDE). KF-STRIDE is focused on improving the ability to express personal strengths during the job interview, a skill that is not taught with VR training. The proposed IMPRESSIVE intervention, which combines the learning of 2 critical abilities (social skills and strength identification), has never been examined in individuals with ASD. Thus, the current proposal will be the first to examine the efficacy of these 2 combined tools in this at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of ASD
* or am a typically developing adolescent
* Able to speak and read English fluently

Exclusion Criteria:

* History of stroke, traumatic brain injury, or any other neurological injury or disease
* History of significant psychiatric illness (bipolar, schizophrenia or psychosis)
* Uncontrolled seizures
* Any other unstable medical complications

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Mock Job Interview Change | 8 weeks
  Mock Job Interview skills will be assessed by having blinded raters trained to assess job interviews scoring participants across a number of domains including expressing personal strengths and sounding professional. This rating scheme has been used in previous research (Smith et al., 2014; 2015),

SECONDARY OUTCOMES:
Self-reported job interview skills | 8 weeks
  Questionnaire to assess self-perceived skills
self-reported job interview anxiety | 8 weeks
  Questionnaire to assess self-perceived anxiety
Employment readiness | 8 weeks
  Questionnaire to assess self-perceived employment readiness
Job Search Behavior | 8 weeks
  Questionnaire to assess self-perceived job search behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Helen Genova, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No